CLINICAL TRIAL: NCT00618111
Title: A Single Dose, 4-Period, 2-Treatment Replicate Design Bioequivalency Study of Granisetron Hydrochloride 1 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GRAN-T1-PVFD-1
Record Dates: First submitted 2008-01-30; First posted 2008-02-18 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Nausea; Vomiting
Keywords: Prevention of nausea and vomiting associated with radiation or chemotherapy
MeSH Terms: conditions — Nausea; Vomiting | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Granisetron

SUMMARY:
The objective of this study was to assess bioequivalence of a potential generic 1 mg granisetron tablet formulation compared with Roche Laboratories' 1 mg granisetron tablet, Kytril, following a single 1 mg dose, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to granisetron or any other comparable or similar product.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2005-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, 4-period, 7 day washout

CONTACTS AND LOCATIONS:
Overall Officials: James Kissling, M.D., Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States